CLINICAL TRIAL: NCT05811442
Title: A Phase IIa, Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of 50561 in Patients With Mild or Moderate Alzheimer's Disease
Brief Title: Study of 50561 in Patients With Mild or Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Joekai Biotechnology LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 50561-II-01
Record Dates: First submitted 2023-03-28; First posted 2023-04-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; 50561; Rac1
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 50561 256mg (Experimental): 50561 at a dose of 256mg n=20 group
  Interventions: Drug: 50561 high dose
- 50561 128mg (Experimental): 50561 at a dose of 128mg n=20 group
  Interventions: Drug: 50561 low dose
- placebo (Placebo Comparator): Placebo n=20 group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 50561 high dose — study drug
  Arms: 50561 256mg
Drug: 50561 low dose — study drug
  Arms: 50561 128mg
Drug: Placebo — Non-active study drug
  Arms: placebo

SUMMARY:
This is a multi-center, Phase IIa, randomized, double-blind, placebo-controlled study designed to evaluate the efficacy, safety of two doses of 50561 compared to placebo in participants diagnosed with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate and sign the informed consent form (ICF) with a legal guardian;
2. Male or female subjects aged 50-85 years (inclusive), at the time of informed consent;
3. Subjects have received education in primary school and above and are able to complete protocol specified cognitive ability test and other tests;
4. Meets the National Institute on Aging -Alzheimer's Association (NIA-AA) core clinical criteria (2011) for probable Alzheimer's disease (AD) dementia;
5. Impaired memory for at least 12 months, with a tendency of progressive aggravation;
6. Treatment-naive subjects for Alzheimer's disease (AD);
7. Mild to moderate Alzheimer's disease (AD):

(1) Mini-Mental State Examination (MMSE) score of ≥ 11 and < 26 (2) Clinical Dementia Rating-Global Score (CDR-GS) of 1 or 2;

8. Hachinski Ischemic Scale (HIS) score of ≤ 4;

9. Hamilton Depression Rating Scale (HAMD) (17-item version) score of ≤ 10;

10. Cranial magnetic resonance imaging (MRI) plain scan and oblique coronal hippocampal scan:

1. Age-adjusted medial temporal lobe atrophy scale [MTA scale] score: Score 2 or more for < 75 years, score 3 or more for ≥ 75 years;
2. Infarction lesions larger than 2 cm in diameter ≤ 2
3. Without infarction lesion in vital sites, such as the thalamus, hippocampus, entorhinal cortex, paraolfactory cortex, angular gyrus, cortex, and other subcortical gray matter nuclei;
4. Fazekas Scale ≤ 2.

11. If female with childbearing potential, tests negative for pregnancy at screening and baseline visits. Male and female patients with childbearing potentials agree to use contraceptives with an annual failure rate of < 1% throughout the trial and for 90 d after the last dose;

12. Subject shall have a stable and reliable caregiver who provides care for at least 2 h per day for 4 d per week. The caregiver must accompany the subject in all visits and have sufficient interaction and communication with the subject in order to assist the investigator in completing the relevant assessments.

Exclusion Criteria:

1. Dementia caused by other reasons: Vascular dementia, central nervous system infection (e.g., AIDS, syphilis), Creutzfeldt-Jakob disease, Huntington's disease, Parkinson's disease, Lewy body dementia, brain trauma dementia, other physical and chemical factors (e.g., drug poisoning, alcohol poisoning, carbon monoxide poisoning), important corporeal diseases (e.g., hepatic encephalopathy, pulmonary encephalopathy), intracranial space-occupying lesions (e.g., subdural hematoma, brain tumors), endocrine system disorders (e.g., thyroid disease, parathyroid disease ) and dementia due to vitamin deficiency or any other known causes;
2. Previously had/currently has nervous system disorder (including Neuromyelitis optica, Parkinson's disease, epilepsy);
3. Mental disorders confirmed according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), including schizophrenia or other mental illness, bipolar disorder, major depression, or delirium;
4. Laboratory test abnormalities at screening visit and baseline: Liver function (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) > 2-fold the upper limit of normal (ULN); Kidney function (creatinine [Cr]) > 1.5-fold the ULN; Creatine kinase (CK) > 2-fold the ULN; Patients with values that slightly exceed these ranges but are not clinically significant may be included as assessed by the investigator;
5. Presence of any one of the following infections at the screening visit:

(1) Positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) and positive for hepatitis B virus deoxyribonucleic acid (HBV-DNA) (exceeding the upper limit of the normal range of the study site); (2) Positive for anti-hepatitis C virus (HCV) antibody (Ab); (3) Positive for human immunodeficiency virus (HIV) Ab; (4) Positive for Treponema pallidum (TP) Ab;

6. Presence of other active and poorly managed systemic bacterial, viral, fungal, or parasitic infections (except for fungal nail infection) at the screening visit, or other clinically significant active infections that render the subject unsuitable for study participation as assessed by the investigator;

7. Systolic blood pressure (SBP) ≥ 160 mmHg or < 90 mmHg or diastolic blood pressure (DBP) ≥ 100 mmHg or < 60 mmHg at the screening visit and baseline; Patients with SBP or DBP that slightly exceed this range but is not clinically significant may be included as assessed by the investigator;

8. Prolonged corrected QTc interval (Fridericia formula, Appendix 14.1) in the 12-lead electrocardiography (ECG) at screening visit and baseline: Fridericia corrected QT interval (QTcF) > 450 ms for males and > 470 ms for females or other clinically significant ECG abnormalities that render the subject unsuitable for study participation (e.g., heart rate < 50 beats/min, sinus node dysfunction, Mobitz II or third-degree atrioventricular block);

9. Patients with unstable or severe cardiovascular, respiratory, digestive, urinary, hematologic, or endocrine disorders within 6 months prior to the screening visit, including pancreatitis, severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, life-threatening ventricular arrhythmia requiring maintenance therapy, pulmonary hypertension, respiratory failure, previous hypoglycemia coma, unstable blood glucose control in diabetic patients, and stroke (including transient ischemic attack), and are unsuitable for study participation as assessed by the investigator;

10. Presence of gastrointestinal disorder that, as assessed by the investigator, can impact drug absorption or metabolism within 6 months prior to the screening visit;

11. Underwent major surgery within 6 months prior to the screening visit that renders the patient unsuitable for enrollment or planning to undergo major surgery during the study;

12. Suffered from a malignant tumor within 3 years prior to the screening visit (excluding resected basal cell carcinoma or cutaneous squamous cell carcinoma , and/or resected carcinoma in situ);

13. Received other traditional Chinese or Western nootropic medications/treatments within 4 weeks prior to baseline;

14. Use of strong CYP3A4 inhibitor or strong CYP3A4 inducer within 4 weeks or 5 half-lives (whichever is longer) prior to baseline;

15. Received other investigational drugs within 4 weeks prior to baseline;

16. Received vaccines within 4 weeks prior to baseline;

17. Alcohol abuse or drug abuse within 1 year prior to the screening visit;

18. History of severe allergy, non-allergic drug reaction or multiple drug allergy, or known history of allergy to 50561 tablet and its excipients;

19. Lacks adequate premorbid literacy, adequate vision, or adequate hearing to complete the required psychometric tests;

20. Breastfeeding women;

21. Other conditions that render the subject unsuitable for study participation as assessed by the investigator.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognition (ADAS-Cog 13) | 24 weeks
  Change from baseline in the Alzheimer's Disease Assessment Scale-Cognition (ADAS-Cog 13) at 24 weeks.
  The total score ranges from 0 to 85, with higher scores representing worse outcome.

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognition (ADAS-Cog 13) | 6 weeks, 12 weeks
  Change from baseline in the Alzheimer's Disease Assessment Scale-Cognition (ADAS-Cog 13) at 6 weeks and 12 weeks. The total score ranges from 0 to 85, with higher scores representing worse outcome.
Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) | 6 weeks, 12 weeks, 24 weeks
  Change from baseline in the Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) scale at 6 weeks, 12 weeks and 24 weeks. The total score ranges from 0 to 18, with higher scores representing worse outcome.
Mini-Mental State Examination (MMSE) | 6 weeks, 12 weeks, 24 weeks
  Change from baseline in the Mini-Mental State Examination (MMSE) at 6 weeks, 12 weeks and 24 weeks. The total score ranges from 0 to 30, with higher scores representing better outcome.
Alzheimer's Disease Collaborative research group-Activities of Daily Living (ADCS-ADL) | 6 weeks, 12 weeks, 24 weeks
  Change from baseline in the Alzheimer's Disease Collaborative research group-Activities of Daily Living (ADCS-ADL) at 6 weeks, 12 weeks and 24 weeks. The total score ranges from 0 to 78, with higher scores representing better outcome.
Neuropsychiatric Inventory (NPI) | 6 weeks, 12 weeks, 24 weeks
  Change from baseline in the 12-item behavioral domain scores on the Neuropsychiatric Inventory (NPI) scale at 6 weeks, 12 weeks and 24 weeks. The total score ranges from 0 to 144, with higher scores representing worse outcome.
Neuropsychiatric Inventory (NPI) | 6 weeks, 12 weeks, 24 weeks
  Change from baseline in the caregiver stress scores on the Neuropsychiatric Inventory (NPI) scale at 6 weeks, 12 weeks and 24 weeks. The total score ranges from 0 to 60, with higher scores representing worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Jia, Principal Investigator — Xuanwu Hospital, Beijing
Locations (12):
- China (12):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Anding Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Heilongjiang Provincial Hospital of Traditional Chinese Medicine, Haerbin, Heilongjiang
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First affiliated hospital of SOOCHOW university, Suzhou, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided